CLINICAL TRIAL: NCT00304616
Title: A Multi-center, Randomized, Open, Treatment-switching Study From Orally Administered Antipsychotic Monotherapy in the Treatment of Chronic Schizophrenic and Schizoaffective Patients
Brief Title: SWitching to Abilify Trial (SWAT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Korea Otsuka Pharmaceutical Co.,Ltd., Korea Otsuka Pharmaceutical Co.,Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOP-010402
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Aripiprazole
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole; Amisulpride; Olanzapine; Quetiapine Fumarate; Risperidone

INTERVENTIONS:
Drug: Aripiprazole, Solian, Olanzapine, Seroquel, Risperidone

SUMMARY:
To evaluate the efficacy, safety and tolerance of an 12 and 26-week aripiprazole administration

DETAILED DESCRIPTION:
This trial was designed to evaluate the efficacy, safety and tolerance of an 12 and 26-week aripiprazole administration to schizophrenic outpatients who maintain stable (no change with dosage, usage, route of the most recent antipsychotic drugs) symptoms and discontinued previous antipsychotic drugs.

Aripiprazole (10~30 mg/day) will be orally administered for 12 weeks followed by an extension phase for a maximum of an additional 14 weeks (total of 26 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Men and women, ages 18 to 65. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized.
* Patients who have not been hospitalized during last three months
* Patients who have kept clinically stable dosage during last one month
* Patients with a diagnosis of schizophrenia and schizoaffective disorder as defined by DSM-IV criteria
* Patients whose symptoms are not optimally controlled or whose antipsychotic medication is not well-tolerated, which in the clinical judgment of the treating psychiatrist require a change of treatment.
* Patients who have received antipsychotics in the past must have shown a response to a neuroleptic medication other than clozapine.

Exclusion Criteria:

* Patients who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period
* Women who are pregnant or breastfeeding
* Patients who are at risk for committing suicide: either having active suicidal ideation considered clinically significant or recently attempted suicide
* Patients with a diagnosis of bipolar disorder, depression with psychotic symptoms, or organic brain syndromes
* Patients who have met DSM-IV criteria for any significant Psychoactive Substance Use Disorder within the 3 months prior to Screening
* Patients considered treatment-resistant to antipsychotic medication (patients need to have shown a previous response to a antipsychotic medication other than clozapine) and patients with a significant history of intolerance to multiple antipsychotic treatments
* Treatment with a long-acting antipsychotic (i.e., haloperidol decanoate or fluphenazine decanoate) in which the last dose was within 3 weeks of randomization.
* Patients with a history of neuroleptic malignant syndrome
* Patients with epilepsy, a history of seizures (except for a single childhood febrile seizure), or a history of an abnormal EEG, severe head trauma, or stroke or who have a history or evidence of other medical conditions (e.g., congestive heart failure) that would expose them to an undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the course of the trial
* Patients who would be likely to require prohibited concomitant therapy during the trial
* Patients who have previously enrolled in an aripiprazole clinical study or who have participated in any clinical trial with an investigational agent within the past month
* Prisoners or subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-10; Primary Completion 2006-06 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
CGI-I mean score(at week 1, 3, 4, 8 & every 4 weeks until week 26)

SECONDARY OUTCOMES:
Changes in PANSS total & PANSS subscore & depression subscore originated from PANSS (at week 4, 8 & every 4 weeks until week 26
IAQ (at week 8)
POM (at week 1, 2, 4, 8)
GAF (at week 8 & end of study)
CGI-S (at week 1, 3, 4, 8 & every 4 weeks until week 26)
AEs, Vital Signs, Weight gain, Prolactin increase, extrapyramidal syndrome, sleep disturbance, Laboratory tests (at week 1, 2, 4, 8 & every 4 weeks until week 26).

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Yoon Kim, Prof., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea